CLINICAL TRIAL: NCT04456400
Title: Enhancing Ultrasound & Photoacoustic for Recognition of Intestinal Abnormalities (EUPHORIA)
Brief Title: Enhancing Ultrasound & Photoacoustic for Recognition of Intestinal Abnormalities
Acronym: EUPHORIA
Status: Terminated | Type: Observational
Why Stopped: The termination is based on a shifted commercial interest of the Sponsor and is not related to any safety grounds.
Sponsor: iThera Medical GmbH (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: cMSOT-2
Record Dates: First submitted 2020-06-19; First posted 2020-07-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: IBD; UC; CD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Endoscopic histology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation cohort: The derivation sub-cohort will be used to derive optimum reconstruction algorithm parameters of MSOT images.
  Primary objective of the derivation cohort is to derive Multispectral Optoacoustic Tomography (MSOT) thresholds maximizing receiver operating characteristic (ROC) to distinguish endoscopic remission from active disease.
  As secondary objective, performance of the Multispectral Optoacoustic Tomography (MSOT) device will be analyzed.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography (MSOT)
- Validation cohort: Objective of the validation cohort is to confirm the performance of Multispectral Optoacoustic Tomography (MSOT) using prescribed thresholds from the derivation cohort.
  Interventions: Diagnostic Test: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Diagnostic Test: Multispectral Optoacoustic Tomography (MSOT) — cMSOT-2 system is indicated for measurement of the Multispectral Optoacoustic Tomography (MSOT) values in the bowel wall of patients with an established diagnosis of inflammatory bowel disease (IBD), specifically Crohn's Disease (CD) and Ulcerative Colitis (UC). The MSOT values provided may be used as an aid to the assessment of inflammatory disease activity in the bowel wall.

SUMMARY:
The clinical investigation aims to generate clinical data to support the use of Multispectral Optoacoustic Tomography (MSOT) in clinical practice, its inclusion in diagnostic guidelines and to support its reimbursement, specifically to

* Further validate the application with respect to including ulcerative colitis patients
* Prepare a study protocol for large-scale clinical validation study in inflammatory bowel disease (IBD)
* Successfully execute the clinical validation study

DETAILED DESCRIPTION:
The clinical investigation, EUPHORIA, will pave the way to establish Multispectral Optoacoustic Tomography (MSOT) technology for the non-invasive assessment of intestinal inflammation in patients. EUPHORIA will enable commercialization of the technology by finalizing technical improvements that will increase diagnostic outcome beyond what has been shown in a first feasibility study, will improve usability, prepare CE marking for the new device and validate clinical results in a large clinical investigation.

Inflammatory bowel disease (IBD) is a chronic condition, posing significant burden to patients and health care systems. Patients suffer from a relapsing course of intestinal inflammation, and to date, there is no satisfying noninvasive diagnostic modality for monitoring disease activity. In a recent clinical study conducted by University Hospital Erlangen, MSOT, a technology developed by iThera Medical (ITM), has proven to be superior in diagnostic performance to other procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of UC or CD for at least three months prior to enrollment
2. Age ≥ 18 years
3. Indication for endoscopy according to institutes routine care
4. Written informed consent

Exclusion Criteria:

1. Stoma independent of localization, ileoanal pouch
2. Prior bowel surgery other than ileocecal resection, which potentially affects the study procedure by fundamentally changing bowel anatomy by removing the ROI (e.g. (partial) resection of the sigmoid, left sided colon) or repositioning the ROI to an inaccessible location (e.g. right-sided colectomy with transversostomy)
3. Indeterminate Colitis, irritable bowel syndrome (IBS)
4. Involvement of the upper gastrointestinal (GI) track only
5. Isolated proctitis
6. Complications, such as infectious enteritis, infectious colitis and infectious enterocolitis, abscess formation, intestinal obstruction, toxic megacolon
7. Tattoo in skin area of interest
8. Skin lesions, scar tissue or skin diseases affecting the area of imaging
9. Highly pigmented skin in the area of imaging (e.g. Fitzpatrick skin type V and VI)
10. The bowel wall is invisible in the Ultrasound image of the MSOT system
11. Medication leading to increased light sensitivity
12. Pregnant and breastfeeding women
13. Mental retardation of the patient with restriction of general judgment and awareness
14. Exclusion due to safety concerns of investigator (subject who has any condition, including any physical, psychological, or psychiatric condition, which in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data and renders the subject an unsuitable candidate for the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of CD or UC in whom endoscopy is indicated
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Derivation Cohort: derive optimum diagnostic MSOT thresholds | 5-10 days
  Derivation cohort: The primary endpoint of the derivation cohort is to derive optimum diagnostic MSOT thresholds based on receiver operating characteristics (ROC) analysis to distinguish endoscopic active disease from remission in Crohn's Disease (CD) or Ulcerative Colitis (UC) patients.
Validation cohort: re-assess the diagnostic accuracy of MSOT | 5-10 days
  Validation cohort:
  The primary endpoint of the validation cohort is to re-assess the diagnostic accuracy of MSOT to distinguish endoscopic active disease from remission in an independent cohort. It will be considered successful if a lower 90% confidence of limit at least 75% of area under curve (AUC) is reached

SECONDARY OUTCOMES:
Derivation Cohort: MSOT thresholds | 9-10 months
  Derive MSOT thresholds using histology as a reference: receiver operating characteristics (ROC) analysis to distinguish histologic active disease from remission.
Derivation Cohort: MSOT performance, diagnostic accuracy measures | 9-10 months
  Diagnostic accuracy measures (area under curve (AUC), sensitivity, specificity) of MSOT to distinguish endoscopic active disease from remission.
Derivation Cohort: MSOT performance, diagnostic accuracy | 9-10 months
  Diagnostic accuracy of MSOT to distinguish histologic active disease from remission
Validation Cohort: MSOT performance, diagnostic accuracy measures | through study completion, an average of 1 year
  Further diagnostic accuracy measures (sensitivity, specificity, predictive values) of MSOT to distinguish endoscopic active disease from remission using the MSOT thresholds from the derivation cohort
Validation Cohort: MSOT performance, diagnostic accuracy | through study completion, an average of 1 year
  Diagnostic accuracy (area under curve (AUC), sensitivity, specificity, predictive values) of MSOT to distinguish histologic active disease from remission using the MSOT thresholds from the derivation cohort.
Both cohorts: diagnostic accuracy | through study completion, an average of 1 year
  Diagnostic accuracy of MSOT to distinguish clinical active disease from remission.
Both cohorts: performance of other non-invasive diagnostic modalities | through study completion, an average of 1 year
  Assess performance of other non-invasive diagnostic modalities in order to allow for comparison to MSOT performance. Diagnostic accuracy of each of the various non-invasive tests (CRP, fCal, US, MRI) with respect to the endoscopy (reference test) and histology will be calculated using standard techniques for diagnostic studies. This includes cross tabulation of the index test results by the results of the reference standard, as well as plots of their distribution and ROC curves. Area under the Curve (AUC) estimates and conﬁdence intervals (DeLong) will be calculated. Score conﬁdence intervals (Wilson) will be calculated for proportions such as sensitivity, speciﬁcity, and predictive values at the predeﬁned thresholds.
Both cohorts: likelihood ratios and predictive values for active inflammation | through study completion, an average of 1 year
  Assess the likelihood ratios and predictive values for active inflammation after MSOT examination.
Both cohorts: performance of MSOT in combination with other modalities | through study completion, an average of 1 year
  Explore performance of MSOT in combination with other modalities, e.g. in combination with ultrasound (US) or laboratory. AUC will be estimated for all non-invasive tests with a 95% conﬁdence interval (DeLong) both from the derivation cohort and from the pooled cohorts (derivation + validation) for increased precision. Cohen's κ will be used as a measure of overall agreement. Results will be presented in three-way tables, comparing the new test (MSOT), the non-reference standard (non-invasive modalities), and the reference standard (endoscopy).
Both cohorts: discriminate different grades of disease activity | through study completion, an average of 1 year
  Investigate ability of MSOT and other non-invasive diagnostic modalities, i.e. ultrasoiund (US), fecal calprotectin (fCal), clinical scores to discriminate different grades of disease activity (remission, mild, moderate, high according to endoscopy, histology or clinical scores; for cut-offs.
Both cohorts: interobserver variability | through study completion, an average of 1 year
  Explore variations in MSOT diagnostic accuracy between sites and operators (interobserver variability).
Both cohorts: patient preference | 5-10 days
  Evaluate patient preference for different tests using a patient survey
Derivation cohort: MSOT thresholds using clinical scores as a reference | through study completion, an average of 1 year
  Derive MSOT thresholds using clinical scores as a reference: ROC analysis to distinguish clinical active disease from remission (only derivation cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Waldner, Prof. Dr., Principal Investigator — Universitätsklinikum Erlangen Medizinische Klinik 1
Locations (6):
- Germany (3):
  - Charité- Universitätsmedizin Berlin, Campus Benjamin Franklin, Klinik für Gastroenterologie, Infektiologie und Rheumatologie, Hindenburgdamm 30, Berlin
  - Universitätsklinikum Erlangen Medizinische Klinik 1, Erlangen
  - Universitätsklinikum Jena, Jena
- Italy (3):
  - Policlinico Tor Vergata, Rome, Lazio
  - Centro per la Ricerca e la Cura delle Malattie Infiammatorie Croniche Intestinali IRCCS Humanitas, Rozzano, Lombardy
  - I.R.C.C.S.San Raffaele, Gastroenterology and Gastrointestinal Endoscopy, Via Olgettina 60, Milan

IPD SHARING:
Plan to Share IPD: Undecided